CLINICAL TRIAL: NCT00588523
Title: A Phase II Trial of Intensive Chemotherapy and Autotransplantation for Patients With Newly Diagnosed Anaplastic Oligodendroglioma
Brief Title: Intensive Chemotherapy and Autotransplantation for Patients With Newly Diagnosed Anaplastic Oligodendroglioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of Calgary (Other); Northwestern University (Other); Northwestern Memorial Hospital (Other); Massachusetts General Hospital (Other); Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-089
Record Dates: First submitted 2007-12-22; First posted 2008-01-08 (Estimated); Results first posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-02

CONDITIONS: CNS Cancer; CNS BRAIN
Keywords: Brain; CNS; TEMOZOLOMIDE; Busulfan; Thiotepa
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Busulfan; Thiotepa

ARMS (1):
- 1 (Experimental): temozolomide followed by high dose busulfan and thiotepa
  Interventions: Drug: temozolomide followed by high dose busulfan and thiotepa

INTERVENTIONS:
Drug: temozolomide followed by high dose busulfan and thiotepa — Temozolomide 200mg/m2 PO Days 1-5 recycled every 28 days Day minus -8 thiotepa 250 mg/m2 intravenously Day minus -7 thiotepa 250 mg/m2 intravenously Day minus -6 thiotepa 250 mg/m2 intravenously Day minus -5 busulfan 3.2 mg/kg intravenously over two hours Day minus -4 busulfan 3.2 mg/kg intravenously over two hours Day minus -3 busulfan 3.2 mg/kg intravenously over two hours Day minus -2 rest Day minus -1 rest Day 0 peripheral blood stem cell or bone marrow reinfusion

SUMMARY:
The purpose of this study is to see how effective treatment of high doses of chemotherapy is for your tumor. We will also be looking at the side effects and risks of this treatment.

You will receive very high doses of chemotherapy. High doses of chemotherapy can destroy tumor cells, but it can also destroy normal bone marrow cells. These cells produce white blood cells (which fight infection), red blood cells (which carry oxygen) and platelets (which allow your blood to clot). With too few of these cells there is a serious risk of infection and bleeding.

Therefore, before treatment begins, we will collect some of your own blood cells, called peripheral blood progenitor cells (PBPCs). These cells help create new blood cells. The PBPCs are frozen and saved while you are being treated. Then at the end of treatment, your PBPCs are thawed and given back to you. These healthy PBPCs will replace the blood cells that the high dose chemotherapy destroys and allow your bone marrow to recover and produce blood cells. In a prior study we treated 69 patients in a similar way. More than half were able to avoid or delay brain radiation. This new study will use a different high dose chemotherapy regimen.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic evidence of an anaplastic oligodendroglioma. For this study, World Health Organization classification criteria will be used. Central pathology review must take place prior to high-dose therapy but need not occur prior to study entry and induction therapy.
* Pathologic evidence of an anaplastic mixed glioma (i.e. oligoastrocytoma). Again, histopathologic diagnosis will be made using World Health Organization classification criteria. To qualify as a mixed tumor there must be a minimum of 25% oligodendroglial element. Central pathology review must take place prior to high-dose therapy but need not occur in advance of enrollment or induction therapy.
* The diagnostic surgical procedure may have been a complete resection, partial resection, or biopsy.
* Karnofsky performance status > or equal to 60.
* Granulocyte count > or equal to 1.5 X 109/L.
* Platelet count > or equal to 100 X 109/L
* SGOT < than or equal to 2X upper limit of normal.
* Serum creatinine < than or equal to 1.5X upper limit of normal
* Bilirubin < than or equal to 1.5X upper limit of normal
* All patients must sign written informed consent.

Exclusion Criteria:

* Systemic or leptomeningeal metastases (excluding contiguous leptomeninges)
* Prior cranial radiotherapy or systemic chemotherapy
* Other concurrent malignancy (with the exception of cervical carcinoma in situ or basal cell carcinoma of the skin) or serious illness if this would interfere with the prescribed treatment.
* Pregnant or lactating women
* Refusal to use effective contraception

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2002-09 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kaley, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Thomas AA, Abrey LE, Terziev R, Raizer J, Martinez NL, Forsyth P, Paleologos N, Matasar M, Sauter CS, Moskowitz C, Nimer SD, DeAngelis LM, Kaley T, Grimm S, Louis DN, Cairncross JG, Panageas KS, Briggs S, Faivre G, Mohile NA, Mehta J, Jonsson P, Chakravarty D, Gao J, Schultz N, Brennan CW, Huse JT, Omuro A. Multicenter phase II study of temozolomide and myeloablative chemotherapy with autologous stem cell transplant for newly diagnosed anaplastic oligodendroglioma. Neuro Oncol. 2017 Oct 1;19(10):1380-1390. doi: 10.1093/neuonc/nox086. PMID 28472509
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Newly Diagnosed Anaplastic Oligodendroglioma: temozolomide followed by high dose busulfan and thiotepa
Period: Overall Study
Arm/Group | Participants With Newly Diagnosed Anaplastic Oligodendroglioma
Started | 60
Completed | 57
Not Completed | 3
Not completed — Not treated | 3

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Newly Diagnosed Anaplastic Oligodendroglioma
Number analyzed (Participants) | 60
Age, Continuous [Median (Full Range); unit: years] | 45 [19 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 57
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 53
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Progession Free Survival
Description: To determine the duration of disease control of newly diagnosed pure and mixed anaplastic oligodendrogliomas treated with dose-intensive chemotherapy requiring hematopoietic stem cell support.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: % of participants without progression
Arm/Group | Participants With Newly Diagnosed Anaplastic Oligodendroglioma
Number analyzed (Participants) | 60
% of participants without progression | 85.7 [62 to 95.2]

2. Secondary Outcome: Number of Participants Evaluated for Toxicities
Time Frame: up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Newly Diagnosed Anaplastic Oligodendroglioma
Number analyzed (Participants) | 60
Participants | 60

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Participants With Newly Diagnosed Anaplastic Oligodendroglioma
All-Cause Mortality (participants affected / at risk) | 30/60
Serious Adverse Events (participants affected / at risk) | 26/60
Other Adverse Events (participants affected / at risk) | 57/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Newly Diagnosed Anaplastic Oligodendroglioma (N=60)
Abdominal cramping (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Bilirubin (Investigations) | 1
CNS Hemorrhage (Blood and lymphatic system disorders) | 1
CNS Necrosis/cystic progression (Nervous system disorders) | 1
Catheter related infection (Infections and infestations) | 1
Colitis (Gastrointestinal disorders) | 1
Confusion (Psychiatric disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Delusions (Psychiatric disorders) | 1
Derm, skin other (Skin and subcutaneous tissue disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Encephalopathy (Nervous system disorders) | 1
Fatigue (General disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 6
Fever (General disorders) | 5
Fracture (Musculoskeletal and connective tissue disorders) | 1
Gastrointestinal, other (Gastrointestinal disorders) | 1
Hematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Pneumonia (Infections and infestations) | 2
Wound infection (Infections and infestations) | 1
Infection unk ANC (Infections and infestations) | 1
Infection w/out neutropenia (Infections and infestations) | 2
Insomnia (Psychiatric disorders) | 1
White blood cells (Investigations) | 1
Liver dysfunction/failure (Hepatobiliary disorders) | 1
Mood alteration/anxiety (Psychiatric disorders) | 1
Muscle weakness - whole body/general (Musculoskeletal and connective tissue disorders) | 2
Nausea (Gastrointestinal disorders) | 5
Neurology, other (Nervous system disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1
Headache (Nervous system disorders) | 2
Pancreatitis (Gastrointestinal disorders) | 1
Platelets (Investigations) | 4
Rash, dequamation (Skin and subcutaneous tissue disorders) | 1
Seizure (Nervous system disorders) | 6
Thrombosis (Vascular disorders) | 1
Veno-Occlusive Disease (Vascular disorders) | 2
Vomiting (Gastrointestinal disorders) | 5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Newly Diagnosed Anaplastic Oligodendroglioma (N=60)
Platelets (Investigations) | 16
Leukocytes (Investigations) | 16
Neutrophils (Investigations) | 13
Fatigue (General disorders) | 12
Hemoglobin (Investigations) | 10
Nausea (Gastrointestinal disorders) | 17
Platelets (Investigations) | 8
Constipation (Gastrointestinal disorders) | 6
Fatigue (General disorders) | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 10
Fever (General disorders) | 5
Vomiting (Gastrointestinal disorders) | 10
Diarrhea (Gastrointestinal disorders) | 7
Edema (General disorders) | 4
Headache (Nervous system disorders) | 4
Lymphopenia (Investigations) | 4
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4
Seizure (Nervous system disorders) | 4
AST, SGOT (Investigations) | 3
Abdominal pain/cramping (Gastrointestinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Fever (General disorders) | 3
Pain - other (General disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-26): https://cdn.clinicaltrials.gov/large-docs/23/NCT00588523/Prot_SAP_000.pdf